CLINICAL TRIAL: NCT01162876
Title: A Clinical Pharmacology Study of Saxagliptin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 262-09-003; JapicCTI-101190 (Other: JAPIC)
Record Dates: First submitted 2010-07-12; First posted 2010-07-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
Keywords: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- saxagliptin (Experimental): 5 mg daily for 14days
  Interventions: Drug: saxaglipitin

INTERVENTIONS:
Drug: saxaglipitin — oral administration of 5 mg tablet before breakfast for 14 consecutive days

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and pharmacodynamics of saxagliptin administered before breakfast for 14 consecutive days in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria will be included:

  1. HbA1c level ≥7.0% and < 9.0%
  2. Fasting glucose level ≥130mg/dL and <210mg/dL
  3. Patients who are capable of giving informed consent
  4. Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner for the entire study period and for 4 weeks after completion of the study

Exclusion Criteria:

* Patients with type 1 diabetes mellitus; patients with diabetes mellitus due to other specified drugs, mechanisms, or diseases; and patients with gestational diabetes mellitus
* Patients with a medical history of diabetic coma
* Patients with heart failure
* Patients with a complication of active chronic hepatitis or hepatic cirrhosis
* Patients undergoing treatment of glomerular diseases other than diabetic nephropathy
* Patients with a history or complication of malignant tumor

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | daily, up to 42days
  Concentrations of plasma saxagliptin and BMS-510849
Pharmacodynamics | daily, up to 42 days
  Plasma DPP4 actyivity Concentrations of blood glucose, C-peptide, insulin and glucagon Plasma active GLP-1 concentration

SECONDARY OUTCOMES:
Safety issues | daily, up to 42 days
  Adverse events, skin symptom findings, blood pressure and pulse rate, body temperature, body weight, hypoglycemic symptoms, 12-lead ECG, clinical laboratory tests, and pregnancy test (in women of childbearing potential only)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyushu Clinical Pharmacology Reserch Clinic, Fukuoka, Japan